CLINICAL TRIAL: NCT06096571
Title: An Open-label, Randomized, Response-adaptive Crossover Study to Investigate the Comparative Pharmacokinetics and Bioequivalence of Aterixen 100 mg Tablets and Aterixen 100 mg Film-coated Tablets in Healthy Volunteers
Brief Title: Pharmacokinetics and Bioequivalence of Aterixen 100 mg Tablets and Aterixen 100 mg Film-coated Tablets in Healthy Volunteers
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Valenta Pharm JSC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: ХС221-05-05-2022
Record Dates: First submitted 2023-10-13; First posted 2023-10-24 (Actual); Last update posted 2024-03-29 (Actual); Status verified 2023-10

CONDITIONS: Viral Infection COVID-19

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental: RT-sequence (Other): Group 1 (18 volunteers, RT sequence) will take 1 tablet of Aterixen,100 mg as a single dose in the fasting state in Period 1 and 1 tablet of Aterixen,100 mg film-coated tablet as a single dose in the fasting conditions in Period 2
  Interventions: Drug: Aterixen
- Experimental: TR-sequence (Other): Group 2 (18 volunteers, TR sequence) will take 1 tablet of Aterixen,100 mg film-coated tablet as a single dose in the fasting state in Period 1 and 1 tablet of Aterixen,100 mg as a single dose in the fasting conditions in Period 2
  Interventions: Drug: Aterixen

INTERVENTIONS:
Drug: Aterixen — A single dose of R or T drug in each of 2 periods of the study in fasted conditions

SUMMARY:
1. Comparative evaluation of the safety of the drug Aterixen 100 mg tablets (Valenta Pharm JSC, Russia) and Aterixen 100 mg film-coated tablets (Valenta Pharm JSC, Russia) administered in single doses under fasting conditions in healthy volunteers, based on AE/SAE (adverse events/serious adverse event) analysis;
2. Comparative assessment of pharmacokinetic parameters and bioavailability of Aterixen 100 mg tablets (Valenta Pharm JSC, Russia) and Aterixen 100 mg film-coated tablets (Valenta Pharm JSC, Russia) administered in single doses under fasting conditions in healthy volunteers.
3. To conclude on the bioequivalence of Aterixen 100 mg tablets (Valenta Pharm JSC, Russia) and Aterixen 100 mg film-coated tablets (Valenta Pharm JSC, Russia) administered in single doses under fasting conditions in healthy volunteers.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntary and handwritten informed consent form signed by a healthy volunteer to participate in the study prior to any of the study procedures;
2. Healthy male and female caucasian volunteers aged 18 to 45 years (inclusive);
3. Verified diagnosis "healthy" (without abnormal findings in the protocol-defined clinical, laboratory, and instrumental test data);
4. Blood pressure (BP) levels: 99 to 129 mm Hg, inclusive (systolic, SBP), 70 to 89 mm Hg, inclusive (diastolic, DBP);
5. Heart rate (HR) of 60 to 89 bpm, inclusive;
6. Respiratory rate (RR) of 12 to 20 breaths per minute, inclusive;
7. Body temperature of 36°C to 36.9°C, inclusive;
8. Body mass index (BMI) of 18.5 kg/m2 ≤ BMI ≤ 30 kg/m2, where the body weight range is ≥ 55 kg for men and ≥ 45 kg for women;
9. Consent to use adequate methods of contraception throughout the study and for 30 days after completion; for women of preserved reproductive potential, a negative urine pregnancy test result.

Exclusion Criteria:

1. A history of allergy;
2. Drug intolerance to the active substance N1-[2-(1-Methyl imidazol-4-yl)-ethyl]perhydroazin-2,6-dione (the active ingredient of Aterixen) and/or excipients contained in the studied drug in the anamnesis;
3. History of drug intolerance of N1-[2-(1-Methyl imidazol-4-yl)-ethyl]perhydroazin-2,6-dione (the active ingredient of Aterixen) aand/or excipients contained in the studied drug in the anamnesis;
4. History of hereditary galactose intolerance, lactase or glucose-galactose malabsorption
5. Chronic diseases of the kidneys, liver, gastrointestinal tract (GIT); disease of the circulatory, lymphatic, respiratory, nervous, endocrine, musculoskeletal, urogenital and the immune systems; dermal, hematopoietic, and ophthalmological diseases;
6. History of gastrointestinal surgery (except appendectomy at least 1 year prior to screening);
7. Diseases/conditions that, in the opinion of the investigator, may affect absorption, distribution, metabolism or excretion of the investigational drugs;
8. Acute infectious disease less than 4 weeks prior to screening;
9. Taking medications that significantly affect hemodynamics and medications that affect liver function (barbiturates, omeprazole, cimetidine, etc.) less than 2 months prior to screening;
10. Regularly taking an medicine less than 2 weeks before screening and taking a single medicine less than 7 days before screening (including OTC medicinal products, vitamins, dietary supplements, or medicinal herbs);
11. Donating blood or plasma less than 3 months before screening;
12. Use of hormonal contraceptives (in women) less than 2 months before screening;
13. The use of depot injections of any drug less than 3 months before screening;
14. Pregnancy or lactation; positive urine pregnancy test for women of preserved reproductive potential;
15. Women of preserved reproductive potential with a history of unprotected intercourse within 30 days prior to study drug administration with an unsterilized partner;
16. Participation in another clinical trial less than 3 months prior to screening or concurrently with the present study;
17. Taking more than 10 units of alcohol (1 unit of alcohol is equivalent to 500 ml of beer, 200 ml of wine or 50 ml of spirits) a week within a month prior to the enrollment in the study or history data of alcohol/drug dependence or drug abuse;
18. Smoking more than 10 cigarettes per day currently, or a history of smoking the specified number of cigarettes during the 6 months prior to screening; disagreement to abstain from smoking for the duration of the hospital stay;
19. Consumption of alcohol, caffeine, and xanthine-containing products 7 days prior to the study drug admission;
20. Consumption of citrus fruits, cranberries and products containing them, preparations or products containing St. John's wort - 7 days before admission to the study drug;
21. Dehydration due to diarrhea, vomiting, or other reason within the last 24 hours prior to study drug administration;
22. Positive blood tests for antibodies to human immunodeficiency virus (HIV) 1 and 2, antibodies to Treponema pallidum antigens, hepatitis B surface antigen (HBsAg), antibodies to hepatitis C virus antigens at screening;
23. Positive rapid test for Coronavirus disease 2019 virus (COVID-19) at screening;
24. Clinically significant abnormalities on an electrocardiogram (ECG) history and/or at screening;
25. Positive urinalysis for narcotics and powerful drugs at screening;
26. Positive breath alcohol vapor test at screening.
27. Scheduling an inpatient stay at the time of the study, for any reason other than hospitalization required by this protocol;
28. Inability or inability to meet the requirements of the protocol, perform the procedures prescribed by the protocol, follow the diet, activity regimen.
29. Belonging to a vulnerable group of volunteers: students of higher and secondary medical, pharmaceutical and dental schools, junior staff of clinics and laboratories, employees of pharmaceutical companies, servicemen and prisoners, persons in nursing homes, low-income and unemployed, national minorities, homeless people, vagrants, refugees, persons under guardianship or custody, and persons unable to give consent, and law enforcement officers;
30. Other conditions that, in the opinion of the Researcher, prevent the inclusion of the volunteer in the study or that might lead to early withdrawal of the volunteer from the study, including fasting or a special diet (e.g. vegetarian, vegan, restricted salt intake) or a special lifestyle (night work, extreme physical activity).

Withdrawal Criteria:

1. The volunteer's refusal to further participate in the study;
2. Failure of the volunteer to comply with the rules of participation in the study (skipping study procedures, independent use of drugs prohibited in the study, violation of dietary and lifestyle restrictions, etc.);
3. Occurrence of causes/occurrence during the study of situations that threaten the safety of the volunteer (e.g., hypersensitivity reactions, etc.);
4. Volunteers selected for the study in violation of the inclusion/inclusion criteria;
5. Development of severe adverse event in the volunteer during the study;
6. The volunteer is undergoing or requires treatment that may affect the pharmacokinetic parameters;
7. Missing 2 or more consecutive blood samples or 3 or more blood samples during the same Study Period;
8. Occurrence of vomiting/diarrhea within 4 hours of study drug administration;
9. Positive urine test for narcotics and powerful drugs;
10. Positive breath alcohol vapor test.
11. Positive pregnancy test in women;
12. Positive test for COVID-19;
13. The occurrence in the course of the study of other reasons that prevent the study according to the protocol.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Estimated)
Dates: Start 2024-06-15 (Estimated); Primary Completion 2024-12-15 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
Pharmacokinetics - Cmax | From 0 to 12 hours (Day 1-2 and Day 8-9)
  Maximum plasma concentration (Cmax)
Pharmacokinetics - tmax | From 0 to 12 hours (Day 1-2 and Day 8-9)
  Time to reach Cmax (tmax)
Pharmacokinetics - AUC0-t | From 0 to 12 hours (Day 1-2 and Day 8-9)
  Area under the plasma concentration-time curve from time 0 to t (AUC0-t)
Pharmacokinetics - AUC0-inf | From 0 to 12 hours (Day 1-2 and Day 8-9)
  Area under the plasma concentration-time curve from time 0 to infinity (AUC0-inf)
Pharmacokinetics - AUCextr | From 0 to 12 hours (Day 1-2 and Day 8-9)
  Extrapolated AUC, area under the concentration-time pharmacokinetic curve, to be calculated as Clast/Kel
Pharmacokinetics - t1/2 | From 0 to 12 hours (Day 1-2 and Day 8-9)
  Elimination half-life (t1/2)
Pharmacokinetics - Kel | From 0 to 12 hours (Day 1-2 and Day 8-9)
  Elimination constant (Kel)
Pharmacokinetics - number of points in terminal logarithmic phase | From 0 to 12 hours (Day 1-2 and Day 8-9)
  Used to estimate Kel
Bioequivalence - ratio of Cmax | From 0 to 12 hours (Day 1-2 and Day 8-9)
  Ratio of geometric mean Cmax after intake of R or T (with 90% confidence intervals)
Bioequivalence - ratio of AUC0-t | From 0 to 12 hours (Day 1-2 and Day 8-9)
  Ratio of geometric mean AUC0-t after intake of R or T (with 90% confidence intervals)
Bioequivalence - ratio of AUC0-inf | From 0 to 12 hours (Day 1-2 and Day 8-9)
  Ratio of geometric mean AUC0-inf after intake of R or T (with 90% confidence intervals)

SECONDARY OUTCOMES:
Safety and Tolerability: adverse event (AE) number and frequency | From the screening (and signing informed consent form) to Day 14 of the study or to an early termination visit within the time frame of the study (from Day 0 to Day 14)
  Number and frequency of adverse events (AEs) or serious AEs (SAEs)
Safety and Tolerability: adverse event (AE) characteristics | From the screening (and signing informed consent form) to Day 14 of the study or to an early termination visit within the time frame of the study (from Day 0 to Day 14)
  Description and severity of AEs or serious AEs (SAEs), concomitant therapy for AEs/SAEs, causal relationship, outcomes.
Safety and Tolerability: vital signs - systolic blood pressure (SBP) | Screening, from Day 0 to Day 2, from Day 7 to Day 9, and/or on early termination visit within the time frame of the study (from Day 0 to Day 14)
  SBP, mmHg
Safety and Tolerability: vital signs - diastolic blood pressure (DBP) | Screening, from Day 0 to Day 2, from Day 7 to Day 9, and/or on early termination visit within the time frame of the study (from Day 0 to Day 14)
  DBP, mmHg
Safety and Tolerability: vital signs - respiratory rate (RR) | Screening, from Day 0 to Day 2, from Day 7 to Day 9, and/or on early termination visit within the time frame of the study (from Day 0 to Day 14)
  RR, breaths per minute
Safety and Tolerability: vital signs - heart rate (HR) | Screening, from Day 0 to Day 2, from Day 7 to Day 9, and/or on early termination visit within the time frame of the study (from Day 0 to Day 14)
  HR, beats per minute
Safety and Tolerability: vital signs - body temperature | Screening, from Day 0 to Day 2, from Day 7 to Day 9, and/or on early termination visit within the time frame of the study (from Day 0 to Day 14)
  Body temperature, centigrade scale
Safety and Tolerability: physical examination results | Screening, from Day 0 to Day 2, from Day 7 to Day 9, and/or on early termination visit within the time frame of the study (from Day 0 to Day 14)
  Number of participants with abnormal physical examination results
Safety and Tolerability: 12-lead electrocardiogram (ECG) - heart rate | Screening, Day 2, Day 9 or on early termination visit within the time frame of the study (from Day 0 to Day 14)
  12-lead ECG (I, II, III, aVR, aVL, aVF, V1-V6) taken while lying down: heart rate (beats per minute)
Safety and Tolerability: 12-lead electrocardiogram (ECG) - PQ interval | Screening, Day 2, Day 9 or on early termination visit within the time frame of the study (from Day 0 to Day 14)
  12-lead ECG (I, II, III, aVR, aVL, aVF, V1-V6) taken while lying down: PQ interval (ms)
Safety and Tolerability: 12-lead electrocardiogram (ECG) - QRS complex | Screening, Day 2, Day 9 or on early termination visit within the time frame of the study (from Day 0 to Day 14)
  12-lead ECG (I, II, III, aVR, aVL, aVF, V1-V6) taken while lying down: QRS complex (ms)
Safety and Tolerability: 12-lead electrocardiogram (ECG) - corrected QT interval (QTc) | Screening, Day 2, Day 9 or on early termination visit within the time frame of the study (from Day 0 to Day 14)
  12-lead ECG (I, II, III, aVR, aVL, aVF, V1-V6) taken while lying down: QTc (ms)
Safety and Tolerability: urinalysis - color | Screening, Day 2, Day 9 or on early termination visit within the time frame of the study (from Day 0 to Day 14)
  Color of the urine
Safety and Tolerability: urinalysis - transparency | Screening, Day 2, Day 9 or on early termination visit within the time frame of the study (from Day 0 to Day 14)
  Transparency of the urine
Safety and Tolerability: urinalysis - pH | Screening, Day 2, Day 9 or on early termination visit within the time frame of the study (from Day 0 to Day 14)
  pH of the urine
Safety and Tolerability: urinalysis - specific gravity | Screening, Day 2, Day 9 or on early termination visit within the time frame of the study (from Day 0 to Day 14)
  Specific gravity of the urine
Safety and Tolerability: urinalysis - protein | Screening, Day 2, Day 9 or on early termination visit within the time frame of the study (from Day 0 to Day 14)
  Protein in the urine (g/L)
Safety and Tolerability: urinalysis - glucose | Screening, Day 2, Day 9 or on early termination visit within the time frame of the study (from Day 0 to Day 14)
  Glucose in the urine (mmol/L)
Safety and Tolerability: urinalysis (microscopy) - red blood cells | Screening, Day 2, Day 9 or on early termination visit within the time frame of the study (from Day 0 to Day 14)
  Red blood cells in the urine (number in sight)
Safety and Tolerability: urinalysis (microscopy) - white blood cells | Screening, Day 2, Day 9 or on early termination visit within the time frame of the study (from Day 0 to Day 14)
  White blood cells in the urine (number in sight)
Safety and Tolerability: urinalysis (microscopy) - epithelial cells | Screening, Day 2, Day 9 or on early termination visit within the time frame of the study (from Day 0 to Day 14)
  Epithelial cells in the urine (number in sight)
Safety and Tolerability: urinalysis (microscopy) - cylinders | Screening, Day 2, Day 9 or on early termination visit within the time frame of the study (from Day 0 to Day 14)
  Cylinders in the urine (number in sight)
Safety and Tolerability: urinalysis (microscopy) - mucus | Screening, Day 2, Day 9 or on early termination visit within the time frame of the study (from Day 0 to Day 14)
  Mucus in the urine (presence in sight)
Safety and Tolerability: urinalysis (microscopy) - bacteria | Screening, Day 2, Day 9 or on early termination visit within the time frame of the study (from Day 0 to Day 14)
  Bacteria in the urine (number in sight)
Safety and Tolerability: complete blood count - hemoglobin | Screening, Day 2, Day 9 or on early termination visit within the time frame of the study (from Day 0 to Day 14)
  Hemoglobin, g/dL
Safety and Tolerability: complete blood count - red blood cells | Screening, Day 2, Day 9 or on early termination visit within the time frame of the study (from Day 0 to Day 14)
  Red blood cells, 10^6/uL
Safety and Tolerability: complete blood count - hematocrit | Screening, Day 2, Day 9 or on early termination visit within the time frame of the study (from Day 0 to Day 14)
  Hematocrit, %
Safety and Tolerability: complete blood count - platelets | Screening, Day 2, Day 9 or on early termination visit within the time frame of the study (from Day 0 to Day 14)
  Platelets, 10^3/uL
Safety and Tolerability: complete blood count - white blood cells | Screening, Day 2, Day 9 or on early termination visit within the time frame of the study (from Day 0 to Day 14)
  White blood cells, 10^3/uL
Safety and Tolerability: complete blood count - erythrocyte sedimentation rate | Screening, Day 2, Day 9 or on early termination visit within the time frame of the study (from Day 0 to Day 14)
  Erythrocyte sedimentation rate, mm per hour
Safety and Tolerability: complete blood count - neutrophils | Screening, Day 2, Day 9 or on early termination visit within the time frame of the study (from Day 0 to Day 14)
  Neutrophils, %
Safety and Tolerability: complete blood count - lymphocytes | Screening, Day 2, Day 9 or on early termination visit within the time frame of the study (from Day 0 to Day 14)
  Lymphocytes, %
Safety and Tolerability: complete blood count - eosinophils | Screening, Day 2, Day 9 or on early termination visit within the time frame of the study (from Day 0 to Day 14)
  Eosinophils, %
Safety and Tolerability: complete blood count - monocytes | Screening, Day 2, Day 9 or on early termination visit within the time frame of the study (from Day 0 to Day 14)
  Monocytes, %
Safety and Tolerability: complete blood count - basophils | Screening, Day 2, Day 9 or on early termination visit within the time frame of the study (from Day 0 to Day 14)
  Basophils, %
Safety and Tolerability: blood test results - total protein | Screening, Day 2, Day 9 or on early termination visit within the time frame of the study (from Day 0 to Day 14)
  Total protein in blood serum, g/L
Safety and Tolerability: blood test results - creatinine | Screening, Day 2, Day 9 or on early termination visit within the time frame of the study (from Day 0 to Day 14)
  Creatinine in blood serum, umol/L
Safety and Tolerability: blood test results - glucose | Screening, Day 2, Day 9 or on early termination visit within the time frame of the study (from Day 0 to Day 14)
  Glucose in blood serum, mmol/L
Safety and Tolerability: blood test results - total bilirubin | Screening, Day 2, Day 9 or on early termination visit within the time frame of the study (from Day 0 to Day 14)
  Total bilirubin in blood serum, umol/L
Safety and Tolerability: blood test results - total cholesterol | Screening, Day 2, Day 9 or on early termination visit within the time frame of the study (from Day 0 to Day 14)
  Total cholesterol in blood serum, mmol/L
Safety and Tolerability: blood test results - alanine transaminase (ALT) | Screening, Day 2, Day 9 or on early termination visit within the time frame of the study (from Day 0 to Day 14)
  ALT in blood serum, U/L
Safety and Tolerability: blood test results - aspartate transaminase (AST) | Screening, Day 2, Day 9 or on early termination visit within the time frame of the study (from Day 0 to Day 14)
  AST in blood serum, U/L
Safety and Tolerability: blood test results - alkaline phosphatase (ALP) | Screening, Day 2, Day 9 or on early termination visit within the time frame of the study (from Day 0 to Day 14)
  ALP in blood serum, U/L

CONTACTS AND LOCATIONS:
Locations (1):
- Limited Liability Company "Research Center Eco-Safety", Saint Petersburg, Russia

IPD SHARING:
Plan to Share IPD: Undecided